CLINICAL TRIAL: NCT00314379
Title: Vitamin E Treatment and Endothelial Function in Type 2 Diabetic Patients With Hp 2-2 Phenotype From the I CARE Study (EFI)
Brief Title: Endothelial Function in a Sample Group of Patients From the ICARE Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Technion, Israel Institute of Technology (Other)
Collaborators: Clalit Health Services (Other); Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HP1980
Record Dates: First submitted 2006-04-10; First posted 2006-04-13 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Cardiovascular Diseases
Keywords: Diabetes; Endothelial Function; Haptoglobin
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus | interventions — Vitamin E

INTERVENTIONS:
Drug: Vitamin E 400IU/day

SUMMARY:
The ICARE study, clinicaltrials.gov ID number: NCT00220831 and protocol number KL-2004, is recruiting diabetic patients with haptoglobin phenotype 2-2, which are randomised to either Vitamin E 400IU per day or placebo. Patients will be followed for 4 years for the major cardiovascular complications of diabetes, acute myocardial infarction (MI), stroke and cardiovascular mortality (see ICARE protocol). The EFI study, Endothelial Function in ICARE will recruit a sample group of 50 patients from the ICARE cohort. These patients will complete all requirements by ICARE protocol and in addition will be tested for endothelial function by a non-invasive method of flow mediated dilatation (FMD).

DETAILED DESCRIPTION:
Fifty patients will be randomly sampled from the ICARE untreated cohort (registry) of diabetic patients with Hp2-2 phenotype which were not randomised to treatment under ICARE study. Patients will be randomised to either vitamin E 400 IU/d or Placebo upon sampling for EFI study.

The patients will be tested for endothelial function by a method of Post Ischemic Flow mediated Dilatation.

all patients will undergo a baseline Endothelial Function test and then start taking the study drug for 2 months. at the end of two months of therapy the patients will undergo a second endothelial function test, then therapy will be stopped for 2 weeks and a cross over will be performed for an additional 2 months of therapy which in the end the third and final endothelial function test will be done.

An interim Results analysis is set to be done once the first 20 patients completed the protocol. In case of significant differences between the groups, study principal investigators will decide about study completion.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients aged 55 and above

Exclusion Criteria:

* Patient who takes antioxidant treatment will be asked to stop, or cannot be included in the study.
* Patients who had a cardiovascular disease (CVD) incident (myocardial infarction [MI], stroke, transient ischemic attack [TIA]), unstable angina pectoris, uncontrolled hypertension (HTN), will have to wait a month after stabilization to be included in the study.
* Allergy to vitamin E.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-04; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function by a non-invasive method of FMD

SECONDARY OUTCOMES:
Predefined in the protocol submitted to the EC approved prior to study beginning and the Inform Consent Form signed by all study participants prior to study related procedures, serum was preserved for the analysis of oxidative and inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Shany Blum, M.D. M.Sc., Principal Investigator — Technion, Israel Institute of Technology; Uzi Milman, M.D., Principal Investigator — Clalit Health Services; Chen Shapira, M.D., Principal Investigator — Clalit Health Services; Giris Jacob, M.D. Ph.D., Principal Investigator — Rambam Health Care Campus; Lior Dayan, M.D. M.Sc., Principal Investigator — Rambam Health Care Campus; Andrew P Levy, M.D. Ph.D., Principal Investigator — Technion, Israel Institute of Technology
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Asleh R, Blum S, Kalet-Litman S, Alshiek J, Miller-Lotan R, Asaf R, Rock W, Aviram M, Milman U, Shapira C, Abassi Z, Levy AP. Correction of HDL dysfunction in individuals with diabetes and the haptoglobin 2-2 genotype. Diabetes. 2008 Oct;57(10):2794-800. doi: 10.2337/db08-0450. Epub 2008 Jul 3. PMID 18599520